CLINICAL TRIAL: NCT05021770
Title: Safety and Efficacy of Orelabrutinib（O） in Combination With Thiotepa（T） in Refractory and Relapsed Primary CNS Lymphoma： A Single-arm, Multicenter Phase Ib/II Study（OT）
Brief Title: Orelabrutinib in Combination With Thiotepa in Refractory and Relapsed Primary CNS Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huiqiang Huang (Other)
Collaborators: Guangdong 999 Brain Hospital (Other)
Responsible Party: Sponsor-Investigator, Huiqiang Huang, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OT
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Refractory and Relapsed Primary CNS Lymphoma; PCNSL; Non Hodgkin Lymphoma
Keywords: PCNSL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — orelabrutinib; Thiotepa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ib (Experimental): Orelabrutinib dose escalation will occur using a standard 3+3 dose-escalation approach to determined the maximum tolerated dose(MTD) of orelabrutinib dose in combined with thiotepa, beginning at dose level I (150 mg daily) and potentially escalating to dose level 2 (200mg) with rules for escalation and de-escalation. If the dose-limiting toxicity is not found, the dose of 200mg will be used for phase II trial (RP2D).
  Orelabrutinib: 150mg or 200mg orally daily. Thiotepa: The dose of thiotepa is fixed as 30 mg/m2 intravenously every 3 weeks (maximum 6 cycle).
  Interventions: Drug: Orelabrutinib; Drug: Thiotepa
- Phase II (Experimental): Participants will receive orelabrutinib and thiotepa at the pre-determined dosage level established in Phase 1b, until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion. The response will be evaluated every 2 cycles.
  Orelabrutinib: RP2D (150 mg or 200 mg qd) Thiotepa:Sintilimab: The dose of thiotepa is fixed as 30 mg/m2 intravenously every 3 weeks (maximum 6 cycle).
  Interventions: Drug: Orelabrutinib; Drug: Thiotepa

INTERVENTIONS:
Drug: Orelabrutinib — 150mg or 200mg orally daily
  Arms: Phase Ib
Drug: Orelabrutinib — RP2D
  Arms: Phase II
Drug: Thiotepa — 30 mg/m2 intravenously every 3 weeks (maximum 6 cycle)

SUMMARY:
The purpose of this study was to investigate the maximum tolerated dose and efficacy of Orelabrutinib combined with Thiotepa in refractory and relapsed primary central nervous system lymphoma (PCNSL).

ELIGIBILITY:
Inclusion Criteria:

1. Men and woman who aged 18 or older on the day of consenting to the study.
2. Participants must be able to understand and willing to sign a written informed consent document.
3. ECOG performance status of 0 to 2.
4. Histologically documented primary central nervous system(CNS) lymphoma.
5. Participants should have evidence of 1 measurable or evaluable enhancing disease on MRI, PET-CT or PET-MRI.
6. Relapsed or refractory disease with at least 1 prior HD-MTX-based therapy.
7. Life expectancy of > 3 months (in the opinion of the investigator).
8. Any non-hematologic toxicity associated with prior treatment should be stable and recovered to ≤ Grade 1 (according to NCI CTCAE V5.0，except for alopecia)
9. Demonstrate adequate organ function as defined below: (all screening labs should be performed within 14 days of treatment initiation)

   * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L, Platelets ≥ 75 x 10^9/L，Hb ≥80 g/L;
   * International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5 times the upper limit of normal;
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal;
   * Serum bilirubin ≤ 1.5 times the upper limit of normal;
   * Creatinine clearance ≥ 60 mL/min calculated by the Cockcroft-Gault formula using actual body weight.
10. Must be able to tolerate MRI/CT/PET-CT/PET-MRI scans and lumbar puncture.
11. Ability to swallow oral medications.
12. Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study.
13. If the disease progresses after radiotherapy, there is no need for washout period;If the tumor responds after radiotherapy, a 6-month washout period is required.
14. First-line treatment with thiotepa-containing regimens is effective, and patients who relapse after more than 1 year can be enrolled.

Exclusion Criteria:

1. The pathological diagnosis was T-cell lymphoma.
2. Prior therapy with a checkpoint inhibitor or BTK inhibitor.
3. Participation in another clinical study with an investigational product during the 12 weeks prior to the first day of study treatment.
4. Participants requires more than 5 mg of dexamethasone daily or the equivalent for control of primary CNS symptoms lasting for more than 5 days within 14 days.
5. Active bleeding within 4 weeks prior to first administration, or ongoing use of anticoagulant/antiplatelet agents, or tendency to bleeding (e.g., esophageal varices at risk for bleeding, locally active ulcerative lesions) or coagulation disorder as considered by the investigator.
6. Has an uncontrolled or significant cardiovascular disease, including (but not limited to) :

   * Any of the following conditions within 6 months prior to initial administration: congestive heart failure (NYHA class III or IV), myocardial infarction, unstable angina, or arrhythmia requiring treatment at the time of screening, left ventricular ejection fraction (LVEF) <50%;
   * Primary or secondary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmic right ventricular cardiomyopathy, restricted cardiomyopathy, undefined cardiomyopathy);
   * Clinical history of prolonged QTc phase, grade II type II atrioventricular block or grade III atrioventricular block or QTc interval (F method) & GT;470 msec (female) or >;480msec (male).
   * Hypertension, which is difficult to control, is not suitable for this study
7. Uncontrolled infections or infections requiring intravenous antimicrobial treatment.
8. Known active infection with hepatitis C virus (HCV)，hepatitis B virus (HBV) or syphilis as determined by serologic tests and/or PCR.
9. History of or positive human immunodeficiency virus (HIV) screen result.
10. Patient underwent major systemic surgery ≤ 6 weeks prior to starting the trial treatment or who has not recovered from the side effects of such surgery, or who plan to have surgery within 2 weeks of the first dose of the study drug.
11. Previous organ transplantation or allogeneic stem cell transplantation.
12. Pregnant or lactating women, or subjects of childbearing age who do not want to use contraception for 180 days from the study period to the end of the study.
13. History of stroke and intracranial hemorrhage within 6 months before the first administration, except intracranial hemorrhage caused by surgical sequelae.
14. Patient with hepatic、renal 、neurological、psychiatric, or endocrine disease , as Investigator's discretion, is too damaged to participate in this study; Patient having other conditions that should exclude it from the trial, as the Investigator's discretion.
15. Alcohol or drug abuse.
16. Allergic to any component of the investigational product.
17. Participants who received live viral vaccination within 4 weeks from enrollment date. Patients are prohibited from receiving live attenuated vaccines, including influenza vaccines, during the study period.
18. Previous CAR-T therapy.
19. PVRL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Part 1 Dose Escalation：The maximum tolerated dose (MTD) | Incidence of dose limiting toxicities (DLTs) up to 21 days
  To determine the maximum tolerated dose (MTD)
Part 2 Dose Expansion：ORR (Investigator-Assessed) | Up to 2 years
  The overall response rate (ORR) including complete response (CR), unconfirmed complete (CRu) and partial response (PR) according to the 2005 Response Criteria of the International Primary CNS Lymphoma Collaborative Group (IPCG)

SECONDARY OUTCOMES:
Part 1 Dose Escalation：Objective response rate (ORR) | Up to 2 years
  The objective response rate (ORR) is defined as the proportion of patients with a best response of CR, CRu or PR
Part 1 Dose Escalation：Compelet response rate (CRR) | Up to 2 years
  The complete response rate (ORR) is defined as the proportion of patients with a best response of CR or CRu
Part 1 Dose Escalation：Duration of overall response (DOR) | Up to 2 years
  The duration of overall response is measured from the time measurement
Part 1 Dose Escalation：Disease control rate (DCR) | Up to 2 years
  The disease control rate (DCR) is defined as the proportion of patients with a best response of CR, CRu, PR or SD
Part 1 Dose Escalation：Progression-free survival (PFS) | Up to 2 years
  The progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first
Part 1 Dose Escalation：Overall survival (OS) | Up to 2 years
  The overall survival (OS) is defined as the duration of time from start of treatment to time of death.
Part 2 Dose Expansion：Compelet response rate (CRR) | Up to 2 years
  The complete response rate (ORR) is defined as the proportion of patients with a best response of CR or CRu
Part 2 Dose Expansion：Duration of overall response (DOR) | Up to 2 years
  The duration of overall response is measured from the time measurement
Part 2 Dose Expansion：Disease control rate (DCR) | Up to 2 years
  The disease control rate (DCR) is defined as the proportion of patients with a best response of CR, CRu, PR or SD
Part 2 Dose Expansion：Progression-free survival (PFS) | Up to 2 years
  The progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first
Part 2 Dose Expansion：Overall survival (OS) | Up to 2 years
  The overall survival (OS) is defined as the duration of time from start of treatment to time of death.
The toxicity profile of the orelabrutinib and thiotepa combination therapy | Up to 2 years
  All subjects who received at least one dose of OT will be included in the safety analysis. Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0.

OTHER OUTCOMES:
Describe the tumor mutation profile by NGS | Up to 2 years
  DNA from tumor tissue and CSF will be sequencing by next generation sequencing (NGS).Identify the PNCSL-related variants and gene expression alterations by NGS.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China